CLINICAL TRIAL: NCT06657092
Title: Ultrasound Guided Erector Spinae Plane Efficacy of Erector Spinae Plane Block for Analgesia in Breast Surgery
Brief Title: Ultrasound Guided Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gözde Gamze Uzun (Other)
Responsible Party: Sponsor-Investigator, Gözde Gamze Uzun, Consultant Anesthesiologist, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kocaeli Univercity
Record Dates: First submitted 2023-02-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-02

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Intervention Model Description: Patients were randomized into two groups, ESPB and control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- erector spinae plane block group (Active Comparator): Single-shot ultrasound (US)-guided ESP block with 20 ml 0.25% bupivacaine at the T4 vertebral level
  Interventions: Procedure: Erector Spinae Plane Block
- control group (Active Comparator): morphine pca to patient
  Interventions: Procedure: Standart therapy

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Single-shot ultrasound (US)-guided ESP block with 20 ml 0.25% bupivacaine ( Marcaine ) at the T4 vertebral level will be performed.
  Other Names: espb group
  Arms: erector spinae plane block group
Procedure: Standart therapy — Postoperative 0.5 mg/kg morphine and 1 gr paracetamol will be admistered intravenously in the operation theatre and intravenous patient controlled analgesia (PCA) will be performed in the plastic surgery ward postoperatively
  Arms: control group

SUMMARY:
Patients were randomized into two groups, ESP and control. Single-shot ultrasound (US)-guided ESP block with 20 ml 0.25% bupivacaine at the T4 vertebral level was performed preoperatively to all patients in the ESP group. The control group received no intervention. Patients in both groups were provided with intravenous patient-controlled analgesia device containing morphine for postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 age
2. Patients who scheduled for bilateral reduction mammoplasty
3. ASA Class I-II

Exclusion Criteria:

1. Coagulopaty

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | Postoperative total opioid consumption in miligrams will be recorded at hour 24
  Patients in both groups will receive opioid in postoperative period. Total opioid consumption in miligrams will be compared

SECONDARY OUTCOMES:
Intraoperative opioid consumption | At the end of the operation
  The amount of remifentanyl administered to patients via intravenous infusion during the operation in micrograms, will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Unıversity, Kocaeli, izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No